CLINICAL TRIAL: NCT03714581
Title: The Efficacy of Intravaginal Laser Therapy in Women With History of Gynecological Cancer Treated With Pelvic Radiotherapy: Double-blind Randomized Placebo-controlled Trial
Brief Title: Laser Therapy Following Radiotherapy for Gynecological Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Themos Grigoriadis, MD, PhD, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 143/21-03-2018
Record Dates: First submitted 2018-10-14; First posted 2018-10-22 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Radiotherapy; Gynecological Cancer; Dyspareunia; Vaginal Dryness
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): Microablative Fractional CO2 Laser Therapy (The parameters that will be used are the following: 1) Power: 30 ή 40 watts, 2) Dwell time:1000μs, 3) Spacing 1000 μm, 4) Depth: SmartStak parameter from 1-3 depending on the treatment status, 5) D-pulse mode.)
  Interventions: Device: Microablative Fractional CO2 Laser Therapy
- Placebo (Placebo Comparator): Placebo therapy (The parameters that will be used are the following: 1) Power: 0.5 watts, 2) Dwell time:1000μs, 3) Spacing 1000 μm, 4) Depth: SmartStak parameter 1, 5) Smart-pulse mode.
  Interventions: Device: Microablative Fractional CO2 Laser Therapy

INTERVENTIONS:
Device: Microablative Fractional CO2 Laser Therapy — 5 laser therapies intravaginally administered will be applied at monthly intervals.
  Other Names: SmartXide2 V2LR, Monalisa Touch, DEKA, Florence, Italy

SUMMARY:
Women with a history of pelvic radiotherapy due to gynecological cancer, will receive laser therapy for the management of genitourinary syndrome of menopause.

ELIGIBILITY:
Inclusion Criteria:

* History of gynecological cancer treated with pelvic radiotherapy
* last radiotherapy >1 year
* women sexually active or willing to resume sexual activity
* symptoms of dyspareunia, vaginal dryness, itching/burning and vaginal bleeding related to sexual intercourse

Exclusion Criteria:

* Relapse of gynecological cancer
* prolapse stage >1
* active genital infection (i.e herpes, vaginitis)
* underlying pathologies that could interfere with patients compliance to the protocol (i.e any psychiatric condition)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 112 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
10-centimeter Visual Analogue Scale assessing intensity of dyspareunia and dryness | Change from baseline at 1 month post-treatment
  It is a straight line with 2 endpoints "0" and "10". Zero defines "no dyspareunia at all" and "no dryness at all" , while 10 "dyspareunia as bad as it could be" and "dryness as bad as it could be". Participants will draw a line at or between the 2 end points. The distance between zero and drawn line will define the intensity of dyspareunia and dryness

SECONDARY OUTCOMES:
3 days voiding diary | Change from baseline at 1 month post-treatment
  Assesses frequency of urination, amount of urine, presence of urgency and/or urinary incontinence and amount of fluid intake
Day-to Day Impact of vaginal aging questionnaire (DIVA) | Change from baseline at 1 month post-treatment
  It includes 4 domains: activities of daily living (5 items), sexual functioning (5 items), emotional well-being (4 items), self-concept and body image (5-items). Each item of each domain could receive values from 0 to 4. Mean scores are calculated on each of the domain scales. Higher scores indicate greater symptom impact
The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ) cervical cancer module (CX24) | Change from baseline Quality of Life questionnaire (QLQ) cervical cancer module (CX24) at 1-month post-treatment
  It includes 4 functional scales (body image, sexual activity, sexual enjoyment, sexual/vaginal functioning) with 9 items and 5 symptoms scales (symptoms experience, lymphedema, peripheral neuropathy, menopausal symptoms and sexual worry) with 15 items. Each item range from 1 to 4. Higher scores in sexual activity and sexual enjoyment indicate better functioning, while higher scores in all other domains indicate higher impact of cervical cancer
Patients Global Impression of Improvement | At 1-month post-treatment
  It is a single item questionnaire assessing the impression of participants following the intervention
International Consultation on Incontinence Questionnaire Short Form/Female Lower Urinary tract Symptoms (ICIQ-FLUTS) | Change from baseline International Consultation on Incontinence Questionnaire Short Form/Female Lower Urinary tract Symptoms (ICIQ-FLUTS) at 1-month post-treatment
  It is a 12-items questionnaire evaluating nocturia, urgency, bladder pain, frequency, hesitancy, straining, intermittency, urinary incontinence (urge, stress and unexplained), frequency of urinary incontinence and nocturnal enuresis. Filling, voiding and incontinence symptoms subscales range from 0 to 15, 0 to 12 and 0 to 20, respectively.
King's Health Questionnaire (KHQ) | Change from baseline King's Health Questionnaire at 1-month post-treatment
  It has 3 sections: 1) general health and overall health related to urinary symptoms with 2 questions, 2) incontinence impact, role limitations, physical limitations, social limitations, personal limitations, emotions, sleep and energy, and severity coping measures with 19 questions and 3) bother or impact of urinary symptoms with 11 questions. Scores of each domain of the 2 sections range from 0 to 100. Scores of the third section range from 0 to 3. Higher scores indicate higher impact of urinary incontinence.
Female Sexual Function Index | Change from baseline Female Sexual Function Index at 1-month post-treatment
  It includes 6 domains assessing sexual functioning (desire, arousal, orgasm, lubrication, satisfaction and pain). Total score is calculated by summing scores of the 5 domains multiplied by certain factors with a minimum value of 2 and maximum 36
Vaginal Maturation Value | Change from baseline Vaginal Maturation Value at 1-month post-treatment
  It is calculated by defining the percentage of superficial, intermediate and parabasal epithelial cells on the vaginal pap smear, following the formula (1x%superficial)+(0.5x%intermediate)+(0x%parabasal). It may receive values from 0 to 100%.It is considered to be an indicator of the estrogenic stimulation, whereas values of 0-49%, 50-64% and 65-100% indicate absent/low, moderate and high estrogenic effect on the vaginal epithelium, respectively.
Vaginal Health Index Score | Change from baseline Vaginal Health Index Score at 1-month post-treatment
  It evaluates vaginal elasticity, fluid volume, ph of vaginal fluid, epithelial integrity and moisture. Each one of these may receive scores from 1 to 5. Total score is calculated by summing the 5 scores ranging from 5 to 25. Higher scores indicate better vaginal status.
Partner Performance Questionnaire | Change from baseline Partner Performance Questionnaire at 1-month post-treatment
  It evaluates aspects of sexual satisfaction of cancer survivors partners

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Athanasiou, Associate Proffesor, Study Director — National and Kapodistrian University of Athens, Greece
Locations (1):
- Urogynecological Unit of Alexandra Hospital, Athens, Greece

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601
- [Derived] Athanasiou S, Pitsouni E, Grigoriadis T, Michailidis G, Tsiveleka A, Rodolakis A, Loutradis D. A study protocol of vaginal laser therapy in gynecological cancer survivors. Climacteric. 2020 Feb;23(1):53-58. doi: 10.1080/13697137.2019.1646720. Epub 2019 Sep 2. PMID 31474161